CLINICAL TRIAL: NCT06223542
Title: A Phase I Study to Investigate the Safety of the Ubiquitin Activating Enzyme Inhibitor TAK-243 in Adult Solid Tumor and Lymphoma Patients
Brief Title: Studying TAK-243 in Patients With Advanced Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-11194; NCI-2022-11194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10299 (Other: National Cancer Institute LAO); 10299 (Other: CTEP)
Record Dates: First submitted 2024-01-24; First posted 2024-01-25 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Indolent Non-Hodgkin Lymphoma; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; TAK-243

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (twice weekly UAE inhibitor TAK-243) (Experimental): Patients receive UAE inhibitor TAK-243 IV on days 1, 4, 8, and 11 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on study, and undergo CT, MRI, and collection of blood throughout the study, and may undergo ECHO as clinically indicated on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Drug: UAE Inhibitor TAK-243
- Arm B (once weekly UAE inhibitor TAK-243) (Experimental): Patients receive UAE inhibitor TAK-243 IV on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on study, and undergo CT, MRI, and collection of blood throughout the study, and may undergo ECHO as clinically indicated on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Drug: UAE Inhibitor TAK-243

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: UAE Inhibitor TAK-243 — Given IV
  Other Names: AOB87172; MLN7243; TAK-243

SUMMARY:
This phase I trial studies the side effects and best dose of ubiquitin-activating enzyme (UAE) inhibitor TAK-243 (TAK-243) in treating patients with a solid tumor that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic) and in patients with lymphoma. TAK-243 is a drug that binds to and inhibits the ubiquitin-activating enzyme, an enzyme that is more active on cancer cells than healthy cells, inhibiting tumor cell proliferation and survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the safety, tolerability, and the recommended phase II dose of UAE inhibitor TAK-243 (TAK-243) administered twice-weekly or once-weekly in patients with advanced solid tumors and lymphomas.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetic (PK) profiles of TAK-243 administered on twice-weekly and once-weekly schedules in patients with advanced solid tumors and lymphomas.

II. To determine the effects of TAK-243 on levels of K48-linked ubiquitination in pre- and post-treatment tumor biopsies.

III. To observe and record anti-tumor activity.

EXPLORATORY OBJECTIVES:

I. To determine the effects of TAK-243 on the endoplasmic reticulum (ER) stress marker CHOP, Mcl-1-Noxa heterodimer formation, and the apoptosis marker cleaved caspase-3 in pre- and post-treatment tumor biopsies II. To evaluate potential associations between TAK-243 activity and tumor genomic alterations or ribonucleic acid (RNA) expression profiles.

III. To preliminarily assess progression-free survival (PFS) and overall survival (OS) for TAK-243 monotherapy in patients with advanced solid tumors and lymphomas.

OUTLINE: This is a dose-escalation study of TAK-243 followed by a dose-expansion study. Patients are assigned to 1 of 2 arms.

ARM A: Patients receive UAE inhibitor TAK-243 intravenously (IV) on days 1, 4, 8, and 11 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on study, and undergo computed tomography (CT), magnetic resonance imaging (MRI), and collection of blood throughout the study, and may undergo echocardiograms (ECHO) as clinically indicated on study.

ARM B: Patients receive UAE inhibitor TAK-243 IV once weekly (QW) on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on study, and undergo CT, MRI, and collection of blood throughout the study, and may undergo ECHO as clinically indicated on study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented advanced or metastatic solid tumors with relapsed or refractory disease who have received standard-of-care or approved therapies known to confer clinical benefit, or patients with aggressive lymphomas who have received ≥ 2 prior lines of lymphoma-directed therapy and who do not have remaining effective treatment options (including transplant). Additionally, patients with indolent lymphomas must meet criteria for treatment.
* Patients must have measurable or evaluable disease
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Hemoglobin >= 9 g/dL (patients may be transfused to achieve this value; elevated indirect bilirubin due to post-transfusion hemolysis is allowed)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x institutional ULN OR =< 5 x institutional upper limit of normal for patients with liver metastases at baseline
* Creatinine =< 1.5 x institutional ULN OR creatinine clearance >= 60 mL/min/1.73 m^2 by Cockcroft-Gault
* Any prior therapy must have been completed >= 4 weeks, or >= 5 half-lives of the prior agent (whichever is shorter) prior to enrollment on protocol. Prior definitive radiation should have been completed >= 4 weeks prior to enrollment; prior palliative radiation should have been completed >= 2 weeks prior to enrollment. Patients must be >= 2 weeks since any investigational agent administered as part of a Phase 0 study (where a sub-therapeutic dose of drug is administered) and should have recovered to grade 1 or baseline from any toxicities
* Female patients who:

  * Are postmenopausal (age-related amenorrhea >= 12 consecutive months or follicle-stimulating hormone > 40 mIU/mL), for at least 1 year before the screening visit, OR
  * Are surgically sterile (i.e., who had undergone hysterectomy or bilateral oophorectomy), OR

If they are of childbearing potential:

* Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), or
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

  * Male patients, even if surgically sterilized (i.e., status postvasectomy), who:
* Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), or
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

  * The effects of TAK-243 on the developing human fetus are unknown. For this reason and because ubiquitin-activating enzyme inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of TAK-243 administration
  * Ability to understand and the willingness to sign a written informed consent document
  * Willingness to provide blood for research purposes
  * For expansion phase patients, willingness to undergo 2 core needle biopsy procedures for research purposes if there is a lesion or lesions amenable to repeat biopsy
  * Patients on anticoagulation therapy are eligible for this study in the absence of anticipated drug-drug interactions (DDI) between the anticoagulation agent and TAK-243. If DDI are anticipated and another anticoagulation agent that is compatible with TAK-243 exists, the patient will be transitioned to this alternative, TAK-243-compatible anticoagulation agent

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Life-threatening illness unrelated to cancer
* Patients with uncontrolled coagulopathy or bleeding disorder
* Known hepatic cirrhosis or severe pre-existing hepatic impairment
* Known cardiopulmonary disease defined as:

  * Unstable angina pectoris;
  * Congestive heart failure (New York Heart Association [NYHA] class III or IV);
  * Myocardial infarction (MI) within 6 months prior to first dose (patients who had ischemic heart disease such as a [acute coronary syndrome (ACS)], MI, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll);
  * Cardiomyopathy
* Clinically significant arrhythmia:

  * History of polymorphic ventricular fibrillation or torsade de pointes,
  * Permanent atrial fibrillation (a fib), defined as continuous a fib for >= 6 months,
  * Persistent a fib, defined as sustained a fib lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening,
  * Grade 3 a fib defined as symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) or ablation, and
  * Patients with paroxysmal a fib or < grade 3 a fib for period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen
* Prolonged rate corrected QT (QTc) interval >= 470 m/sec, calculated according to institutional guidelines
* Uncontrolled high blood pressure (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg)
* Known moderate to severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis
* Major surgery within 14 days before the first dose of any study drug
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s)
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s)
* Patients with known brain metastases or carcinomatous meningitis are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for >= 1 month after treatment of the brain metastases. Patients on anti-seizure medications may be enrolled at the discretion of the principal investigator
* TAK-243 is primarily metabolized by CYP3A4/5. Therefore, the concomitant use of strong inhibitors of CYP3A4/5 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir and saquinavir) and strong inducers of CYP3A4/5 (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) is not permitted from 14 days prior to enrollment until the end of the study

  * TAK-243 is a substrate for both organic anion transporting polypeptides (OATP) in human hepatocytes and the drug efflux transporter BCRP (ABCG2). Therefore, concomitant use of drugs that are strong inhibitors of BCRP or OATP is not permitted from 14 days prior to enrollment until the end of the study
  * Other medications that are prohibited while on TAK-243 treatment include herbal medications/preparations (except for vitamins). Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of
  * As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients undergoing vaccination with live vaccines and live attenuated vaccines in the 30 days prior to receiving TAK-243, during the study, and for 100 days after the last dose of study drug. Inactivated vaccines are permitted
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAK-243
* Patients with evidence of chronic hepatitis B virus (HBV) infection who are currently on treatment are eligible if they have an undetectable HBV viral load
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Known human immunodeficiency virus (HIV)-positive patients who meet the following criteria will be considered eligible:

  * CD4 count > 350 cells/mm^3
  * Undetectable viral load for 6 months prior to enrollment
  * Maintained on modern therapeutic regimens utilizing non-CYP-interactive agents
  * No history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections
* Pregnant and lactating/breast-feeding women are excluded from this study because TAK-243 is a UAE-inhibiting agent with the potential for teratogenic or abortifacient effects and there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TAK-243

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Within the first cycle of treatment (Arm A: 21-day cycle; Arm B: 28-day cycle)
  The MTD for each arm will be based on the assessment of dose-limiting toxicities (DLTs) and will be defined as the dose level at which less than one-third of patients (< 2/6 patients) treated at that dose experience a DLT, with the next higher dose level demonstrating a one-third or greater number of patients (>= 2/3 or >= 2/6 patients) having DLT.
Recommended phase 2 dose | Within the first cycle of treatment (Arm A: 21-day cycle; Arm B: 28-day cycle)
Incidence of DLTs | Within the first cycle of treatment (Arm A: 21-day cycle; Arm B: 28-day cycle)
  A DLT is defined as an adverse event that is felt to be related (possibly, probably, or definitely) to administration of study drugs, and meets pre-specified criteria. All toxicities will be reported for all patients who receive any amount of study drug on this study.

SECONDARY OUTCOMES:
Pharmacodynamic (PD) variables | Up to 30 days after the last dose of treatment
  With 10 PD sample pairs, there is 90% power to detect a treatment effect equivalent to 1.8 standard deviations (associated with the inter-patient baseline variability of the PD marker) with the paired 2-sample t-test, at the 1-sided .01 significance level (to accommodate multiple endpoints while maintaining a reasonable over-all type 1 error bound), for a given PD variable of interest. PD variables may be log-transformed to achieve more nearly normal distributions.
Objective tumor response | Up to 30 days after the last dose of treatment
  For each of the two administration schedule arms, the objective tumor response rate will be estimated for the entire patient population in a descriptive fashion, including a 2-sided 90% confidence interval.

OTHER OUTCOMES:
Progression-free survival | Up to 30 days after the last dose of treatment
Overall survival | Up to 30 days after the last dose of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Shin, MD, Principal Investigator — National Cancer Institute LAO
Locations (1):
- National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm